Statistical Analysis Plan: SAINT

# **CLINICAL TRIAL STATISTICAL ANALYSIS PLAN**

**Code: SAINT** 

Title of trial: Pilot study to evaluate the potential of ivermectin to reduce

**COVID-19 transmission** 

Phase: IIa

Date of statistical analysis plan: 5 of October 2020 - Version 1.0

**EudraCT number: 2020-001474-29** 

Sponsor: Clínica Universidad de Navarra

Written by: Aina Casellas, ISGlobal

Principal Investigator: Dr. Carlos Chaccour

Clínica Universidad de Navarra

CONFIDENTIAL MAY NOT BE USED, DIVULGED OR PUBLISHED WITHOUT TRIAL SPONSOR'S CONSENT.

Version 1.0  5 of October 2020

## **Approval Page**

EUDRACT No.: 2020-001474-29

The signatures below confirm that the signatories have reviewed and approved this document which shall govern the stipulated statistical analysis tasks of the specified research study.

| Aina Casellas | Head of Statistics |
|---|---|
| Name | Designation |
| $\bigcirc$ | |
| | 5 of October 2020 |
| Signature | Date |
| Sergi Sanz | Reviewer |
| Name | Designation |
| A TOP OF THE PROPERTY OF THE P | |
| 4-1/ | 5 of October 2020 |
| Signature | Date |
| Carlos Chaccour | Approver |
| Name // / / / / / | Designation |
| Valor Vaur | |
| James 1 les | 5 of October 2020 |
| Signature | Date |

## 1 Table of Contents

| 1 | Tab | le of | Contents | 3 |
|---|---|---|---|---|
| 2 | Abb | revia | tions and Definitions | 5 |
| 3 | Intr | oduc | tion | 5 |
| | 3.1 | Pref | face | 5 |
| | 3.2 | Pur | pose of the analyses | 6 |
| 4 | Stud | dy Ob | ejectives and Endpoints | 6 |
| | 4.1 | | n Study Objective | |
| | 4.2 | Sec | ondary Study Objectives | 6 |
| | 4.3 | End | points | 6 |
| | 4.3. | 1 | Primary | 6 |
| | 4.3. | 2 | Secondary | 6 |
| 5 | Stud | dy Me | ethods | 7 |
| | 5.1 | | neral Study Design and Plan | |
| | 5.2 | Equ | ivalence or Non-Inferiority Studies | 7 |
| | 5.3 | Incl | usion-Exclusion Criteria and General Study Population | 8 |
| | 5.3. | 1 | Inclusion criteria | 8 |
| | 5.3. | 2 | Exclusion criteria | |
| | 5.3. | 3 | Criteria for withdrawal | 9 |
| | 5.4 | Ran | domisation and Blinding | 9 |
| | 5.5 | Stud | dy Variables | 9 |
| | 5.5. | 1 | Baseline information (day 1) | 10 |
| | 5.5. | 2 | Previous medical history (day 1) | 10 |
| | 5.5. | 3 | Visit information | 11 |
| | 5.5. | 4 | Concomitant medication (during follow up) | 15 |
| | 5.5. | 5 | Adverse Events (during follow up) | 15 |
| 6 | Sam | iple S | iize | 18 |
| 7 | Gen | eral | Considerations | 19 |
| | 7.1 | Tim | ing of Analyses | 19 |
| | 7.1. | 1 | Full Analysis Population | 19 |
| | 7.1. | 2 | Safety Population | 19 |
| | 7.2 | Cov | ariates and Subgroups | 19 |
| | 7.3 | | sing Data | |
| ١, | orcion 1 | 1 0 | Dags 2 of 21 | F of Octobor 2020 |

| | 7.4 | Multiple Testing | 19 |
|---|---|---|---|
| 8 | Su | mmary of Study Data | 19 |
| | 8.1 | Subject Disposition | 20 |
| | 8.2 | Derived variables | 21 |
| | 8.3 | Concurrent Illnesses and Medical Conditions | 21 |
| | 8.4 | Prior and Concurrent Medications | 21 |
| | 8.5 | Treatment Compliance | |
| 9 | Eff | ficacy Analyses | 21 |
| | 9.1 | Primary Efficacy Analysis | 21 |
| | 9.2 | Secondary Efficacy Analyses | 22 |
| 10 | ) | Safety Analyses | 22 |
| | 10.1 | Extent of Exposure | |
| | 10.2 | Adverse Events | 22 |
| | 10.3 | Deaths, Serious Adverse Events and other Significant Adverse Events | 22 |
| | 10.4 | Pregnancies | 22 |
| | 10.5 | Clinical Laboratory Evaluations | 22 |
| 1: | 1 | Pharmacokinetics | 23 |
| 12 | 2 | Reporting Conventions | 23 |
| 13 | 3 | Technical Details | 23 |
| 14 | 4 | References | 24 |
| 15 | 5 | Listing of Tables, Listings and Figures | 25 |
| | 15.1 | Tables | 25 |
| | 15.2 | Listings | 29 |
| | 15.3 | Figures | 30 |

#### 2 Abbreviations and Definitions

| AE | Adverse Event |
|------|--------------------------------|
| ВМІ | Body Mass Index |
| CI | Confidence interval |
| CRF | Case Report Form |
| Ct | Cycle threshold |
| CUN | Clínica Universidad de Navarra |
| ENT | Ear, Nose, Throat |
| FU | Follow-up |
| LFU | Lost to follow-up |
| mITT | Modified Intention to treat |
| NTDs | Neglected tropical diseases |
| PP | Per Protocol |
| RR | Relative risk ratio |
| RRP | Reports reported by patients |
| SAE | Severe Adverse Event |
| SAP | Statistical Analysis Plan |

#### 3 Introduction

#### 3.1 Preface

As of May 8, 2020, there were a more than 4 million cases of COVID-19 and more than 270,000 deaths worldwide. There is currently no proven treatment for this disease, so drug-based strategies to control COVID-19 are urgently needed. Among the potential approaches to be considered for COVID-19 are early treatment of patients to reduce progression to severe disease, treatment to block or reduce transmission with a drug that reduces viral excretion in the airway, prophylaxis or combinations of either. These strategies could significantly relieve pressure on the health system and decrease indirect deaths due to other diseases requiring intensive care.

Ivermectin is a widely used anti-parasitic drug for the treatment and control of neglected tropical diseases (NTDs) which has shown an excellent safety profile, with more than 2.5 billion doses distributed in the last 30 years. Based on previous evidence, ivermectin could be active against COVID-19 by inhibiting the replication of the virus or by having immunomodulatory effects.


Statistical Analysis Plan: SAINT

#### 3.2 Purpose of the analyses

These analyses will assess the efficacy and safety of ivermectin as a treatment for COVID-19 patients to reduce virus spread.

### 4 Study Objectives and Endpoints

### 4.1 Main Study Objective

To determine the efficacy of a single dose of ivermectin, administered to low risk, non-severe COVID-19 patients in the first 48 hours after symptoms onset to reduce the proportion of patients with detectable SARS-CoV-2 RNA by PCR from nasopharyngeal swab at day seven post-treatment.

### 4.2 Secondary Study Objectives

- 1. To assess the efficacy of ivermectin to reduce the SARS-CoV-2 viral load in the nasopharyngeal swab at day seven post treatment
- 2. To assess the efficacy of ivermectin to improve symptom progression in treated patients
- 3. To assess the proportion of seroconversions at day 21 in treated patients
- 4. To assess the safety of ivermectin at the proposed dose
- 5. To determine the magnitude of immune response against SARS-CoV-2
- 6. To assess the early kinetics of immunity against SARS-CoV-2

### 4.3 Endpoints

### 4.3.1 Primary

Proportion of patients with a positive SARS-CoV-2 PCR from a nasopharyngeal swab at day 7 post-treatment.

#### 4.3.2 Secondary

- 1. Mean viral load as determined by PCR cycle threshold (Ct) at baseline and on days 4, 7, 14 and 21
- 2. Proportion of patients with fever and cough at days 4, 7, 14 and 21 as well as proportion of patients progressing to severe disease or death during the trial.
- 3. Proportion of patients with seroconversion at day 21.
- 4. Proportion of drug-related adverse events during the trial.
- 5. Median levels of IgG, IgM, IgA measured by Luminex, frequencies of innate and SARS-CoV-2-specific T cells assessed by flow cytometry, median levels of inflammatory and activation markers measured by Luminex and transcriptomics.
- 6. Median kinetics of IgG, IgM, IgA levels till day 28.

The analysis of objectives 5 and 6 will be addressed in a supplementary SAP.


## 5 Study Methods

### 5.1 General Study Design and Plan

The SAINT trial is a single center, randomized, double-blind, placebo-controlled, parallel arm, superiority clinical trial.

Participants will be randomized to receive a single dose of 400 mcg/kg ivermectin or a placebo equivalent and followed up for 28 days.

A final study visit will be made for participants who withdraw prematurely from the study or are withdrawn by the investigator. A summary of the study visits and procedures is provided in **Table 1.** Visit Procedures below.

| | Recruitment<br>Day 1 | <b>Visit 2</b><br>Day 4 | Visit 3 Day 7 | <b>Visit 4</b><br>Day 14 | Visit 5<br>Day 21 | <b>Final visit</b><br>Day 28 |
|---|---|---|---|---|---|---|
| Informed consent# | X | | | | | |
| Randomization | X | | | | | |
| Clinical data collection | X | Х | Х | Х | Х | Х |
| Physical examination | Х | Х | Х | Х | Х | Х |
| Laboratory test* | Х | | Х | Х | | |
| Urine pregnancy test | Х | | | | | |
| Nasopharyngeal swab (PCR for SARS-CoV-2) | Х | Х | Х | Х | Х | |
| Serology for SARS-CoV-2 | Х | Х | Х | Х | Х | Х |
| Proinflammatory and activation markers | Х | Х | Х | Х | Х | Х |
| Cell responses (PBMC) | Х | | Х | | | Х |
| Chest x-ray | Х | | | | | |
| Administration of IP | Х | | | | | |
| Daily self-assessment of symptoms | X | | | | | X |
| Evaluation of adverse events | X | | | | | X |
| | • | | | | | |

<sup>#</sup> verbal consent initially, in writing when isolation is concluded

Table 1. Visit Procedures

### **5.2** Equivalence or Non-Inferiority Studies

Not Applicable

<sup>\*</sup> C reactive protein, Procalcitonin, Renal function: urea, creatinine, electrolytes, FBC, Troponin T, CPK, DD, LDH

Statistical Analysis Plan: SAINT

### 5.3 Inclusion-Exclusion Criteria and General Study Population

#### 5.3.1 Inclusion criteria

- Patients diagnosed with COVID-19 in the emergency room of the Clínica Universidad de Navarra with a positive SARS-CoV-2 PCR.
- Residents of the Pamplona basin ("Cuenca de Pamplona")
- The patient should be between the ages of 18 and 60 years
- Negative pregnancy test for women of child bearing age\*
- The patient or his/her representative have given consent to participate in the study.
- The patient should, in the investigator's opinion, be able to comply with all the requirements of the clinical trial (including home follow up during isolation)

\*Women of child bearing age may participate if they use a safe contraceptive method for the entire period of the study and at least one month afterwards. A woman is considered to not have childbearing capacity if she is post-menopausal (minimum of 2 years without menstruation) or has undergone surgical sterilization (at least one month before the study).

#### 5.3.2 Exclusion criteria

- Known history of Ivermectin allergy
- Hypersensitivity to any component of Stromectol<sup>®</sup>
- COVID-19 Pneumonia
  - Diagnosed by the attending physician
  - Identified in a chest X-ray
- Fever or cough present for more than 72 hours
- Positive IgG against SARS-CoV-2 by rapid test
- Age under 18 or over 60 years
- The following co-morbidities (or any other disease that might interfere with the study in the eyes of the investigator):
  - Immunosuppression
  - Chronic Obstructive Pulmonary Disease
  - Diabetes
  - Hypertension
  - Obesity
  - Acute or chronic renal failure
  - History of coronary disease
  - History of cerebrovascular disease
  - Current neoplasm
- Recent travel history to countries that are endemic for Loa loa (Angola, Cameroon, Central African Republic, Chad, Democratic Republic of Congo, Ethiopia, Equatorial, Guinea, Gabon, Republic of Congo, Nigeria and Sudan)
- Current use of CYP 3A4 or P-gp inhibitor drugs such as quinidine, amiodarone, diltiazem, spironolactone, verapamil, clarithromycin, erythromycin, itraconazole, ketoconazole, cyclosporine, tacrolimus, indinavir, ritonavir or cobicistat. Use of critical CYP3A4 substrate drugs such as warfarin.


Statistical Analysis Plan: SAINT

#### 5.3.3 Criteria for withdrawal

Patients will be informed that they may be withdrawn from the study at any time without providing any explanation. Withdrawal may also take place for any of the following reasons:

- Adverse reaction that puts the patient's life at risk, according the principal investigator's judgment.
- Decision made by the patient or the legally authorized person.
- Documented progression of the disease requiring hospitalization in a different center.
- The patient cannot complete the trial visits due to unforeseen circumstances.
- Development of other disorders that, in the opinion of the investigator and in the patient's best interest, make it advisable for him/her to leave the study.
- Administration of treatment with a non-permitted drug.
- The investigator believes that the patient may benefit from a different treatment.
- Loss of monitoring

The investigator shall strive to ensure that the patient agrees to the final trial visit. The data of the withdrawn patients shall be collected up to this final visit. If the withdrawal is the outcome of a Serious adverse event related to ivermectin or SARS-CoV-2, the data shall be collected until the patient recovers or stabilizes.

The subjects shall be replaced if the withdrawal is for a reason different from lack of efficacy of the treatment or appearance of adverse events. All efforts will be made to maintain the total number of assessable patients as per the protocol.

The withdrawal shall be documented in the patient's clinical history, giving the reasons for the decision. A final trial visit should be conducted by the clinical team if possible.

#### 5.4 Randomisation and Blinding

Participants will be randomized to receive a single dose of 400 mcg/kg ivermectin or a placebo equivalent. The randomization code will be generated by the trial statistician using blocks of four individuals that ensure balance between the groups. This randomization will be performed with the module *ralloc* [1] for Stata software [2]. A study identification code with the format "SAINT-##" (##: from 01 to 24) will be generated using a sequence of random numbers so that the randomization number does not match the subject identifier.

The sequence and code used will be kept in an encrypted file accessible only to the trial statistician. A physical copy will be kept on a locked cabinet at the CUN, accessible only to the staff administering the drug who will not enroll or attend to patient care.

This is a double-blind study; the participants and the clinical team will be blinded. The placebo will not be visibly identical, but it will be administered by a researcher not involved in the clinical care or participant follow up.

#### 5.5 Study Variables

The list of variables collected at each study timepoint is provided in the following subsections.


All study visits must be on the planned days, so no visits out of the specified visit days (1, 4, 7, 14, 21 and 28) will be taken into account in the analysis.

### 5.5.1 Baseline information (day 1)

The variables listed below will be assessed on the first visit.

| Variable name | Description | Data type | Coding or |
|---|---|---|---|
| | • | , , | range |
| Demographics | | | |
| Age | Age (years) | Integer | 18-60 |
| Sex | Gender | Integer | 1: Female |
| | | | 2: Male |
| V1_VSHeight | Height (in m) | Real | 1.2-2.2 |
| V1_VSWeight | Weight (in kg) | Real | 40-100 |
| V1_VSBMI | BMI (in kg/m²) | Real | 18-30 |
| Smoking habits an | d alcohol consumption | | |
| Smoke | Smoker or tobacco products user | Integer | 0: No |
| | | | 1: Yes |
| Cigarettes | Number of cigarettes per day | Integer | 0-40 |
| SmokeYears | Smoking duration (in years) | Integer | ?? |
| Alcohol | Alcohol consumption | Integer | 0: No |
| | | | 1: Yes |
| AlcoholUnits | Weekly alcohol consumption (in units) | Integer | 0-20 |
| Medication | Medication | | |
| MedicationTaken | Taking medication | Integer | 0: No |
| | | | 1: Yes |

### 5.5.2 Previous medical history (day 1)

For each preexisting medical condition, the list of variables given below will be collected.

| Variable name | Description | Data<br>type | Coding or range |
|---|---|---|---|
| RELEVANT_HISTORY_MEDICAL | Relevant History Medical | Integer | 0: Other |
| | | | 1: Cardiovascular |
| | | | 2: Respiratory |
| | | | 3: Hepato-biliary |
| | | | 4: Gastro-intestinal |
| | | | 5: Genito-urinary |
| | | | 6: Endocrine |
| | | | 7: Hematological |
| | | | 8: Musculo-skeletal |
| | | | 9: Neoplasia |
| | | | 10: Neurological |
| | | | 11: Psychological |


Sponsor: Clínica Universidad de Navarra

Statistical Analysis Plan: SAINT

| | | | 12: Immunological |
|-----------|--------------------------|---------|----------------------|
| | | | 13: Dermatological |
| | | | 14: Allergies |
| | | | 15: Eyes, ear, nose, |
| | | | throat |
| Details | Details (Diagnosis / | String | |
| | Procedure) | | |
| StartDate | Start Date | Date | |
| Ongoing | Is the medical condition | Integer | 0: No |
| | ongoing? | | 1: Yes |
| EndDate | End Date | Date | |

#### **5.5.3** Visit information

The list below contains those variables assessed recurrently during follow up. Note that not all variables are collected every visit. A superscript indicating the days when the information is collected is provided for those variables not collected at every study visit.

| Variable name | Description | Data<br>type | Coding or range |
|---|---|---|---|
| VIVisitDate | Visit Date | Date | |
| ASAnySymptoms | Does the patient have any of | Integer | 0: No |
| | the symptoms suggestive of COVID-19? | | 1: Yes |
| ASAnyNewSymptoms | Does the patient have any | Integer | 0: No |
| | new symptom suggestive of COVID-19? | | 1: Yes |
| SYMPTOM | Symptom | Integer | 1: General |
| | | | 2: ENT |
| | | | 3: Respiratory |
| | | | 4: Digestive |
| | | | 5: Other |
| VSHeartRate | Heart rate (beats per minute) | Integer | 50-120 |
| VSBloodPressSystolic | Systolic blood pressure (mmHg) | Integer | 90-160 |
| VSBloodPressDiastolic | Diastolic blood pressure (mmHg) | Integer | 50-100 |
| VSTemperature | Temperature (ºC) | Real | 35-41 |
| VSOxygenSaturation | Oxygen saturation (%) | Real | 85- |
| VSRespiratoryRate | Respiratory rate (breaths per minute) | Integer | 8-24 |
| VSHeight | Height (m) | Real | 1.2-2.2 |
| VSWeight | Weight (kg) | Real | 40-100 |
| VSBMI | BMI (kg/m <sup>2</sup> ) | Real | 18-30 |

Sponsor: Clínica Universidad de Navarra

| DHE A ny A bnormal Dhy Evam | Doos the nationt show any | Intogor | 0: No |
|---|---|---|---|
| | Does the patient show any | Integer | |
| | abnormal signs on physical | | 1: Yes |
| | examination? | | |
| · | Does the patient show any | Integer | 0: No |
| | new abnormal signs on | | 1: Yes |
| | physical examination? | | |
| Xray <sup>1</sup> | X-RAY Result | Integer | 0: Normal |
| | | | 1: Abnormal |
| ChestXrayDescription <sup>1</sup> | X-RAY Description: | String | |
| PregnancyTestConducted <sup>1</sup> | Was a pregnancy test | Integer | 0: No |
| | conducted? | | 1: Yes |
| | | | 2: NA |
| PregnancyTestResult 1 | Pregnancy test result | Integer | 0: Negative |
| | | | 1: Positive |
| PCRSwabResults 1,4,7,14,21 | Swab result | Integer | 0: Negative |
| | | | 1: Positive |
| RSCompleteSelfAssessment | Did the participant complete | Integer | 0: No |
| 47449499 | the self-assessment daily | | 1: Yes |
| | since the last visit? | | |
| | Did the participant report any | Integer | 0: No |
| • | negative changes? | | 1: Yes |
| | Did the participant report any | Integer | 0: No |
| , , , | new medications? | integer | 1: Yes |
| Nasopharyngeal swab (PCR for SA | | | 1. 103 |
| | Gene N (PCR sample) – Result | Integer | 1: Detected |
| remen_gen_iv | delle iv (i elv sample) - ivesuit | Integer | 2: Not detected |
| | | | 3: Not detected |
| DCDDCD must be CT N | Cara N (DCD agraphs) Ct | Deel | |
| PCRPCR_muestra_CT_N | Gene N (PCR sample) – Ct | Real | 12-40 (41 if not |
| | | | detected) |
| | Gene N (PCR sample) – | Integer | 0-10 <sup>12</sup> |
| | Quantity (Copies/ml) | | |
| PCRPCR_gen_E | Gene E (PCR sample) – Result | Integer | 1: Detected |
| | | | 2: Not detected |
| | | | 3: Not done |
| PCRPCR_muestra_CT_E | Cono F (DCD comple) Ct | Real | 12-40 (41 if not |
| | Gene E (PCR sample) – Ct | Real | 0 ( |
| 37_33.112_0.2 | Gene E (PCR Sample) – Ct | Neai | detected) |
| | Gene E (PCR sample) – Ct Gene E (PCR sample) – | Integer | , |
| PCRPCR_muestra_Q_E | | | detected) |
| PCRPCR_muestra_Q_E | Gene E (PCR sample) – | | detected) |
| PCRPCR_muestra_Q_E PCRPCR_gen_ab1 | Gene E (PCR sample) –<br>Quantity (Copies/ml) | Integer | detected) 0-10 <sup>12</sup> |
| PCRPCR_muestra_Q_E PCRPCR_gen_ab1 | Gene E (PCR sample) –<br>Quantity (Copies/ml)<br>Gene ab1 (PCR sample) – | Integer | detected) 0-10 <sup>12</sup> 1: Detected |

| | | | detected) |
|---|---|---|---|
| PCRPCR muestra Q ab1 | Gene ab1 (PCR sample) – | Integer | 0-10 <sup>12</sup> |
| FCKFCK_IIIdestra_Q_ab1 | Quantity (Copies/ml) | integer | 0-10 |
| PCRPCR cul N | Gene N (PCR culture) – Result | Integer | 1: Detected |
| FCKFCK_Cdi_N | Gene iv (FCN culture) – Nesuit | integer | 2: Not detected |
| | | | 3: Not detected |
| PCRPCR_cultivo_CT_N | Gene N (PCR culture) – Ct | Real | 12-40 (41 if not |
| PCKPCK_CUITIVO_CI_IN | Gene N (PCN culture) – Ct | Real | detected) |
| PCRPCR_cultivo_Q_N | Gene N (PCR culture) – | Integer | 0-10 <sup>12</sup> |
| FCRFCR_CUITIVO_Q_IV | Quantity (Copies/ml) | integer | 0-10 |
| DCDDCD cul E | Gene E (PCR culture) – Result | Integer | 1: Detected |
| PCRPCR_cul_E | Gene E (PCK culture) – Result | Integer | 2: Not detected |
| | | | 3: Not detected |
| PCRPCR cultivo CT E | Gene E (PCR culture) – Ct | Dool | 12-40 (41 if not |
| PCRPCR_CUITIVO_CI_E | Gene E (PCR culture) – Ct | Real | detected) |
| DCDDCD sulting O F | Gene E (PCR culture) – | Intogor | 0-10 <sup>12</sup> |
| PCRPCR_cultivo_Q_E | , | Integer | 0-10 |
| DCDDCD and also | Quantity (Copies/ml) | Intern | 1. Datastad |
| PCRPCR_cul_ab1 | Gene ab1 (PCR culture) – | Integer | 1: Detected |
| | Result | | 2: Not detected |
| DODDOD III OT III | 6 14 (969 1) 3 | | 3: Not done |
| PCRPCR_cultivo_CT_ab1 | Gene ab1 (PCR culture) – Ct | Real | 12-40 (41 if not |
| | | | detected) |
| PCRPCR_cultivo_Q_ab1 | Gene ab1 (PCR culture) – | Integer | 0-10 <sup>12</sup> |
| 1 ab august august 17.14 | Quantity (Copies/ml) | | |
| Laboratory test 1,7,14 | | Daal | Mala: 0.7.1.2 |
| DIOCHEN ACCEPTAGE | | Real | Male: 0.7-1.2 |
| BIOCHEMCreatinine | Blood creatinine (mg/dL) | 1.1 | Female: 0.5-0.9 |
| BIOCHEMUreaBlood | Urea blood (mg/dL) | Integer | 16.6-48.5 |
| BIOCHEMMDRD | MDRD (mL/min/1.73m <sup>2</sup> ) | Real | 60- |
| BIOCHEMLDH | LDH (UI/L) | Real | 135-225 |
| BIOCHEMCRP | CRP (mg/dL) | Real | 0-0.5 |
| BIOCHEMTroponin | Troponin T (ng/L) | Real | 0-13 |
| BIOCHEMProcalcitonin | Procalcitonin (ng/mL) | Real | 0-0.5 |
| BIOCHEMSodium | Sodium (mEq/L) | Real | 136-145 |
| BIOCHEMPotassium | Potassium (mEq/L) | Real | 3.5-5 |
| BIOCHEMChlorine | Chlorine (mEq/L) | Real | 98-107 |
| BIOCHEMBicarbonate | Bicarbonate (mEq/L) | Real | 22-29 |
| BIOCHEMRemAnion | Remaining anion (mEq/L) | Real | 8-16 |
| | | Real | Male: 30-400 |
| BIOCHEMFerritin | Ferritin (ng/mL) | | Female: 15-150 |
| ВІОСНЕМСРК | CPK (UI/L) | Real | Male: 0-190 |

| | | | Female: 0-170 |
|---|---|---|---|
| BIOCHEMIL6 | IL-6 (pg/mL) | Real | 0-7 |
| COAGDimero | D-Dimer (ng/mL) | Real | 150-500 |
| | | Real | Male: 4.7-5.1 |
| BCRBC | Red blood cells (10 <sup>12</sup> /L) | | Female: 4.2-5.4 |
| | | Real | Male: 14-17 |
| BCHb | Haemoglobin (g/dL) | | Female: 12-16 |
| | | Real | Male: 42-49 |
| BCHto | Hto (%) | | Female: 37-48 |
| BCVCM | VCM (fL) | Real | 80-95 |
| BCHCM | HCM (pg) | Real | 27-31 |
| ВССМНС | CMHC (g/dL) | Real | 33-35 |
| BCRDW | RDW (%) | Real | 11.5-14.5 |
| BCPlaquetas | Platelets (10 <sup>9</sup> /L) | Integer | 150-450 |
| BCVPM | VPM (f/L) | Real | 7.2-11.1 |
| BCPDW | PDW (%) | Real | 25-65 |
| ВСРТС | PTC (%) | Real | 0.12-0.36 |
| BCWBC | White blood cells (10 <sup>9</sup> /L) | Real | 4.8-10.8 |
| BCNeutrophils | Neutrophils (%) | Real | 45-75 |
| BCTotalNeutrophils | Total Neutrophils (10 <sup>9</sup> /L) | Real | 1.5-6.5 |
| BCLymphocytes | Lymphocytes (%) | Real | 20-50 |
| BCTotalLymphocytes | Total Lymphocytes (10 <sup>9</sup> /L) | Real | 1.2-4 |
| BCMonocytes | Monocytes (%) | Real | 2-9 |
| BCTotalMonocytes | Total Monocytes (10 <sup>9</sup> /L) | Real | 0.4-0.8 |
| BCEosinophils | Eosinophils (%) | Real | 0-6 |
| BCTotalEosinophils | Total Eosinophils (10 <sup>9</sup> /L) | Real | 0-0.4 |
| BCBasophils | Basophils (%) | Real | 0-4 |
| BCTotalBasophils | Total Basophils (10 <sup>9</sup> /L) | Real | 0-0.2 |
| Serology | | | |
| SEROLOGYSerSarsCoV2 1,21 | SARS-CoV-2 (COVID-19) | Integer | 0: Negative |
| | Serology result | | 1: Positive |
| BIOBANKEDTA5 | EDTA 5 Biobank collected | Integer | 0: No |
| | | | 1: Yes |
| BIOBANKEDTA5_PBMC | EDTA 5 Biobank (PBMC) | Integer | 0: No |
| | collected | | 1: Yes |
| BIOBANKSerumBiobank | Serum 10 Biobank collected | Integer | 0: No |
| | | | 1: Yes |
| BIOBANKHeparinBiobank | Heparin 10 Biobank collected | Integer | 0: No |
| | | | 1: Yes |

Statistical Analysis Plan: SAINT

Superscripts indicate the days in which each variable is collected. Variables with no superscripts are collected at all visits.

ENT: Ear, Nose, Throat.

### 5.5.4 Concomitant medication (during follow up)

Details on concomitant treatments will be collected during the study.

| Variable name | Description | Data<br>type | Coding or range |
|---|---|---|---|
| Medication | Medication | String | |
| Units | Units | String | |
| FREQ | Frequency | String | |
| TotalDailyDose | Todal daily dose | Integer | |
| Reason | Reason | String | |
| StartDate | Start Date | Date | |
| EndDate | End Date | Date | |
| CMContinuing | Continuing at end of trial? | Integer | 0: No |
| | | | 1: Yes |

### 5.5.5 Adverse Events (during follow up)

For each Adverse Event occurred, the following details will be recorded.

| Variable name | Variable name Description | | Coding or range |
|---|---|---|---|
| AF | Adverse Event name | type | |
| AL | Adverse Event name | String | |
| ChautData | Chart Data | Data | |
| StartDate | Start Date | Date | |
| TimeStart | Start Time | Date | |
| Ongoing | Is the Adverse Event ongoing? | Integer | 0: No |
| | | | 1: Yes |
| EndDate | End Date | Date | |
| TimeEnd | End Time | Date | |
| Outcome | Outcome | Integer | 1: Recovered |
| | | | 2: Recovered with sequelae |
| | | | 3: Continuing |
| | | | 4: Patient Died |
| | | | 5: Change in AE |
| | | | 6: unknown |
| Severity | Severity | Integer | 1: Mild |
| | | | 2: Moderate |
| | | | 3: Severe |
| RelationshipStudyDrug <sup>1</sup> | Plausible relationship to Study | Integer | 0: No |
| | Drug | | 1: Yes |
| ActionTaken | Action taken with Study Drug | Integer | 1: None |


| | | | 2: Dose Reduction |
|---|---|---|---|
| | | | Temporarily |
| | | | 3: Dose Reduced |
| | | | 4: Discontinued Temporarily |
| WithdrawnDueAE | Withdrawn due to an adverse | Integer | 0: No |
| | event? | | 1: Yes |
| SAE | Serious adverse event (SAE)? | Integer | 0: No |
| | | | 1: Yes |
| SAEReporting | If SAE does it require | Integer | 0: No |
| | immediate reporting? | | 1: Yes |

<sup>1:</sup> An event will be considered as related to the study drug if it appears within 5 days after its administration.

### 5.5.6 Daily self-assessment of symptoms

Each patient will give information on the variables below each day during follow up.

| Variable name | Description Data type | | Coding or range |
|---|---|---|---|
| day | Follow up day | Integer | 1-28 |
| como_se_encuentra | How do you fell today? | Integer | 1: Better than yesterday |
| | | | 2: Same as yesterday |
| | | | 3: Worse than yesterday |
| malestar_si_no | Are you feeling generally unwell | Integer | 0: No |
| | or tired? | | 1: Yes |
| malestar_mejor | If feeling generally unwell or tired, | Integer | 1: Better than yesterday |
| | is it: | | 2: Same as yesterday |
| | | | 3: Worse than yesterday |
| temp_si_no | Have you taken your body | Integer | 0: No |
| | temperature? | | 1: Yes |
| temp | What has been your highest | Real | 35-41 |
| | temperature since yesterday? (in | | |
| | ºC) | | |
| fiebre | Have you had a fever since | Integer | 0: No |
| | yesterday? | | 1: Yes |
| tos_si_no | Do you have a cough? | Integer | 0: No |
| | | | 1: Yes |
| tos_es | Your cough is: | Integer | 1: Dry |
| | | | 2: Productive |
| tos_expectoracion | Your expectoration: | Integer | 1: Is whitish |
| | | | 2: Is yellowish |
| | | | 3: Is greenish |
| | | | 4: Has blood |

| tos_esta | Your cough is: | Integer | 1: Better than yesterday |
|---|---|---|---|
| 103_6314 | Tour coughts. | integer | 2: Same as yesterday |
| | | | , , |
| too ooto | Description of the section of difficult | Intono | 3: Worse than yesterday |
| tos_esta | Does your cough make it difficult | Integer | 0: No |
| | for you to eat, drink or talk? | | 1: Yes |
| olores | Can you perceive odours well? | Integer | 0: No |
| | | | 1: Yes |
| mal_sabor | Do you have a bad taste in your | Integer | 0: No |
| | mouth? | | 1: Yes |
| cefalea | Cephalea | Integer | 0: No |
| | | | 1: Yes |
| dolor_cabeza | Do you have a headache? | Integer | 0: No |
| | | | 1: Yes |
| dolor_garganta | Do you have a sore throat? | Integer | 0: No |
| | | | 1: Yes |
| congestion_si_no | Do you have a stuffy nose? | Integer | 0: No |
| | | | 1: Yes |
| fatiga_si_no | Do you have fatigue? (Shortness | Integer | 0: No |
| | of breath?) | | 1: Yes |
| fatiga | You are fatigated: (multiple | Integer | 1: Resting |
| | choice) | | 2: When talking |
| | | | 3: When walking |
| | | | 4: When climbing stairs |
| vomitos_si_no | Do you have vomiting? | Integer | 0: No |
| | Je yea mare remaining. | | 1: Yes |
| casados_por_tos | Is it caused by coughing? | Integer | 0: No |
| casaacs_poi_tes | is it coused by coughing. | intege. | 1: Yes |
| veces_vomitado | How many times have you | Integer | 1- |
| veces_voinitado | vomited since yesterday? | integer | <b>1</b> - |
| diarrea si no | Do you have diarrhea? | Integer | 0: No |
| diarrea_si_rio | bo you have diarrilea: | integer | 1: Yes |
| donosisionos | How many bowel movements | Intogor | 1- |
| deposiciones | · · | Integer | 1- |
| | have you had since yesterday? | 1.1 | 0.01 |
| medicacion_si_no | Have you taken any medication | Integer | 0: No |
| | for these symptoms in the last 24 | | 1: Yes |
| | hours? | | |
| medicacion_cual | If yes, which one? | String | |
| sintomas_1 | Since yesterday, have you | Integer | 1: Confusion / difficulty |
| | experienced any of these | | concentrating on something |
| | symptoms? (multiple choice) | | 2: Dizziness |
| | | | 3: Drowsiness |
| | | | 4: Vertigo |

Sponsor: Clínica Universidad de Navarra

Statistical Analysis Plan: SAINT

| | | | 5: Tremors |
|---|---|---|---|
| sintomas_2 | Since yesterday, have you | Integer | 1: Blurry vision |
| | experienced any of these | | 2: Difficulty focusing on |
| | symptoms? (multiple choice) | | objects or reading |
| | | | 3: Tunnel vision |
| | | | 4: Abnormal colors or shapes |
| | | 5: Blind spots | |
| | | | 6: Floating points |
| sintomas_3 | Since yesterday, have you | Integer | 1: Pruritus (itching) |
| | experienced any of these | | 2: Rash |
| | symptoms? (multiple choice) | | |

### 6 Sample Size

The study will enroll 24 participants, 12 per arm. The sample size has been calculated for comparing two proportions. This sample provides 80% power at 5% significance level using Fisher's unilateral test to determine a difference of 45% (100% vs 55%) in the proportion of participants with positive PCR at day 7. This includes up to one participant lost to follow up (LFU) per arm. We estimated this low LFU level given that the patients will be isolated at home and will have a low risk of progression to severe disease. The 100% positivity rate at day seven is based on the clinical experience at the Clínica Universidad de Navarra. **Figure 1** provides the relationship power-outcome measure for the full sample and one scenario considering LFU of up to two patients per arm.



**Figure 1** Trial power scenarios for different effect size and loss to follow up levels.


Statistical Analysis Plan: SAINT

#### 7 General Considerations

### 7.1 Timing of Analyses

Data will be collected using the ShareCRF platform [3], which uses automatic rules to provide high quality data. No additional cleaning process will be needed. Daily self-assessment of symptoms will be recorded by each participant in an ODK platform. The final analysis will take place after all subjects have completed the final visit or dropped out and after the finalization and approval of this SAP document.

#### 7.1.1 Full Analysis Population

The efficacy analysis will be done per protocol (PP), including all randomized participants for whom there is a PCR result at day seven.

#### 7.1.2 Safety Population

The safety analysis will be done using a modified intention to treat (mITT) approach considering all randomized and treated participants.

#### 7.2 Covariates and Subgroups

No covariate nor subgroup analyses planned.

#### 7.3 Missing Data

All the available data on safety and efficacy shall be included in the data lists and tables. No values shall be allocated for unavailable data.

Any confusing or incorrect data shall be examined in accordance with the standardized data control procedures.

In the analysis of the records reported by patients (RRP), the omitted data shall be allocated by using the last observation carried forward. The omitted standard shall be examined before any allocation. If the omitted standard is clearly informative, the repercussion of the non-random data shall be evaluated using sensitivity analysis.

For the RRP analysis, if a section of subscale from several is missing, the average of the remaining sections shall be used as a scoring scale, as long as at least half of the sections of the scale is available.

#### 7.4 Multiple Testing

Adjustment for multiple testing will not be necessary as there is only one primary outcome.

### 8 Summary of Study Data

Descriptive analyses will use frequency and percentage (based on the non-missing sample size) for qualitative variables and median, interquartile range and n (non-missing sample size) for quantitative variables. Summary tables will be structured using one column per study arm and overall in the order: Placebo, Ivermectin, All subjects.


### 8.1 Subject Disposition

The number of subjects reaching each study stage will be defined as:

- Assessed for eligibility if any information available on section "screening failures" in the baseline visit CRF.
- Randomized if study identifier given and recorded in the baseline visit CRF.
- Reached visit 2, 3, 4, 5 or final if any information available on the CRF corresponding to that visit.
- Analyzed if PCR result at day 7.

A skeleton CONSORT flow diagram is provided below.




Statistical Analysis Plan: SAINT

#### 8.2 Derived variables

The following table contains the list of derived variables that will be used in the analysis.

| Variable name | Description | Calculation | Data | Coding |
|---|---|---|---|---|
| variable flaffic | Description | Calculation | type | or range |
| any_symptom | Any symptom reported | General OR ENT OR Respiratory OR Digestive OR Others | Integer | 0: No<br>1: Yes |
| platelet_lymphocyte | Platelet-Lymphocyte index | Platelet / Lymphocyte | Real | 0- |
| neutrophil_lymphocyte | Neutrophil-<br>Lymphocyte index | Neutrophil / Lymphocyte | Real | 0- |
| severity_pred | Severity predictor | N/L*CRP*D-dimer | Real | 0- |
| vload_change | Viral load change | (viral load [n] – viral load [1]) / viral load [1] | Real | - |
| A list of variables with prefix "vk" | Primary parameters of viral kinetic | Individual curve fits and non-<br>linear mixed effects models | Real | - |

#### 8.3 Concurrent Illnesses and Medical Conditions

No standard coding system will be used for concurrent illnesses and medical conditions. Each condition will be classified according to the affected system (Cardiovascular, Respiratory, Hepato-biliary, Gastro-intestinal, Genito-urinary, Endocrine, Hematological, Musculo-skeletal, Neoplasia, Neurological, Psychological, Immunological, Dermatological, Allergies, "Eyes, ear, nose, throat" or Other). The summary statistics will be produced in accordance to section 7.

#### 8.4 Prior and Concurrent Medications

No standard coding system will be used for medications. The summary statistics will be produced in accordance to section 7.

#### 8.5 Treatment Compliance

Study treatment is administered using the directly observed therapy (DOT) method. With this method, treatment adherence is ensured as a health care professional watches the study participants while they take their medication.

No treatment compliance measures will be calculated.

## 9 Efficacy Analyses

#### 9.1 Primary Efficacy Analysis

The proportion of participants with positive PCR at day seven post treatment will be calculated. Proportions will be compared between study arms using Fisher's exact test and presented as a relative risk ratio (RR), or reduction of the RR (1- RR) if RR lower than 1, and 95% Confidence


Statistical Analysis Plan: SAINT

Interval (CI). Differences will be considered statistically significant if the p-value obtained is lower than 0.05.

### 9.2 Secondary Efficacy Analyses

Secondary endpoints will be analyzed using descriptive methods as explained in section 8. Graphics such as alluvial diagrams and boxplots will be also employed to assess evolution along follow up for qualitative and quantitative variables, respectively. For each symptom and for all as a composite outcome, Kaplan-Meyer survival curves will be used to show time to improvement. The effect of study treatment on the presence of symptoms will be estimated using mixed effect logistic regression models with subject as a random intercept. These models, will be adjusted by day of follow up as symptoms are expected to disappear over time.

We will attempt to fit viral load profiles as quantified by rt-PCR to standard viral kinetics models (e.g. target cell limited models or eclipse models). Fitting strategies will comprise individual curve fits and non-linear mixed effects models. For successful fits, primary parameters of viral kinetic can be derived and compared between treatment arms. Examples include virion clearance rate, cell death rate, cellular infectivity, and acquired immune effects. Given sufficient data, secondary parameters such as peak viral load, time to peak viral load, and exposure as quantified by area under the curve can be calculated.

### 10 Safety Analyses

All the adverse events that occur during the study will be included in the data lists and sorted by patient and order of occurrence. Events that are considered to be related to the treatment (possibly, probably or definitely related to it) will also be included in a table. A table will with the list the adverse events according to maximum intensity will be provided. The deaths and serious adverse events will also be classified in a separate table.

Summary statistics on the number of observed events and their relatedness with the study drug will be presented by study arm and overall.

#### 10.1 Extent of Exposure

The summary statistics will be produced in accordance to section 7.

#### 10.2 Adverse Events

The summary statistics will be produced in accordance to section 7.

#### 10.3 Deaths, Serious Adverse Events and other Significant Adverse Events

The summary statistics will be produced in accordance to section 7.

### 10.4 Pregnancies

Pregnant women will not be included in the trial. Pregnancy tests will be administered before recruitment to all women of child bearing age.

#### **10.5 Clinical Laboratory Evaluations**


The summary statistics will be produced in accordance to section 7.

### 11 Pharmacokinetics

Not applicable.

### 12 Reporting Conventions

P-values greater or equal to 0.001 will be reported to 3 decimal places. P-values less than 0.001 will be reported as '<0.001'. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data.

### 13 Technical Details

The analyses will be conducted using Stata version 16 [2]. Graphs will be produced using the packages *ggplot2* [4] and *ggalluvial* [5] for R version 4.0.2. [6]. The operating system of the computer will be Windows 10.


### 14 References

- [1] P. Ryan, *RALLOC: Stata module to design randomized controlled trials,* revised 28 Jan 2018 ed., Statistical Software Components S319901, Boston College Department of Economics, 1997.
- [2] StataCorp, Stata Statistical Software: Release 16, College Station, TX: StataCorp LLC, 2019.
- [3] "ShareCRF," [Online]. Available: www.ShareCRF.com.
- [4] H. Wickham, ggplot2: Elegant Graphics for Data Analysis, Springer-Verlag New York, 2016.
- [5] J. C. Brunson, ggalluvial: Alluvial Plots in 'ggplot2', 2020.
- [6] R Core Team, R: A Language and Environment for Statistical Computing, Vienna, Austria: R Foundation for Statistical Computing, 2020.


# 15 Listing of Tables, Listings and Figures

### 15.1 Tables

**Table 1**. Baseline description of study participants

| Mariahla | Stud | ly arm | AII - 1-11- |
|---|---|---|---|
| Variable | Placebo | Ivermectin | All subjects |
| Demographics | | | |
| Gender: female <sup>1</sup> | | | |
| Age <sup>2</sup> | | | |
| Height (in m) <sup>2</sup> | | | |
| Weight (in kg) <sup>2</sup> | | | |
| BMI (in kg/m <sup>2</sup> ) <sup>2</sup> | | | |
| Smoking habits and alcohol consumption | | | |
| Smoker or tobacco products user <sup>1</sup> | | | |
| Number of cigarettes per day <sup>2</sup> | | | |
| Smoking duration (in years) <sup>2</sup> | | | |
| Alcohol consumption <sup>1</sup> | | | |
| Weekly alcohol consumption (in units) <sup>2</sup> | | | |
| Medication | | | |
| Taking medication <sup>1, 3</sup> | | | |
| Previous medical history | | | |
| Cardiovascular <sup>1</sup> | | | |
| Respiratory <sup>1</sup> | | | |
| Hepato-biliary <sup>1</sup> | | | |
| Gastro-intestinal <sup>1</sup> | | | |
| Genito-urinary <sup>1</sup> | | | |
| Endocrine <sup>1</sup> | | | |
| Hematological <sup>1</sup> | | | |
| Musculo-skeletal <sup>1</sup> | | | |
| Neoplasia <sup>1</sup> | | | |
| Neurological <sup>1</sup> | | | |
| Psychological <sup>1</sup> | | | |
| Immunological <sup>1</sup> | _ | | |
| Dermatological <sup>1</sup> | | | |
| Allergies <sup>1</sup> | _ | | |
| Eyes, ear, nose, throat <sup>1</sup> | | | |
| Others <sup>1</sup> | _ | | |

<sup>1:</sup> n/N (Percentage)


<sup>2:</sup> Median (IQR) [n]

<sup>3:</sup> includes OTC, vitamins and supplements

 Table 2. Baseline clinical description of study participants

| | | Stud | Study arm | |
|---|---|---|---|---|
| Variable | | Placebo | Ivermectin | All subjects |
| Symptoms | | | | |
| General 1, 3 | | | | |
| ENT <sup>1,4</sup> | | | | |
| Respiratory <sup>1</sup> | | | | |
| Digestive <sup>1</sup> | | | | |
| Others <sup>1</sup> | | | | |
| Physical examination result | s, system affected | 1 | | |
| General appearance <sup>1</sup> | | | | |
| Heart <sup>1</sup> | | | | |
| Lungs <sup>1</sup> | | | | |
| Abdomen <sup>1</sup> | | | | |
| Extremities <sup>1</sup> | | | | |
| Others <sup>1</sup> | | | | |
| Vital signs | | | | 1 |
| Heart rate (in bmp) <sup>2</sup> | | | | |
| Blood pressure (in mmHg) | Systolic <sup>2</sup> | | | |
| | Diastolic <sup>2</sup> | | | |
| Temperature (in ºC) <sup>2</sup> | | | | |
| Oxygen saturation (in %) 2 | | | | |
| Respiratory rate (in breaths | per minute) <sup>2</sup> | | | |
| Chest X-Ray | | | 1 | |
| Abnormal result <sup>1</sup> | | | | |
| Pregnancy test | | 1 | 1 | |
| Test conducted 1,5 | | | | |
| Positive test result 1 | | | | |
| Laboratory results | | 1 | 1 | |
| Positive nasopharyngeal swa | b for SARS-CoV-2 1 | | | |
| Positive for IgG antibodies <sup>1</sup> | | | | |
| IgG antibodies (in mg/dL) <sup>2</sup> | | | | |
| Positive for IgM antibodies <sup>1</sup> | | | | |
| IgM antibodies (in mg/dL) <sup>2</sup> | | | | |
| Positive for IgA antibodies <sup>1</sup> | | | | |
| IgA antibodies (in mg/dL) <sup>2</sup> | | | | |
| Blood creatinine (in mg/dL) | 2 | | | |
| Urea blood <sup>2</sup> | | | | |
| MDRD <sup>2</sup> | | | | |
| LDH (in U/L) <sup>2</sup> | | | | |
| CRP (in mg/L) <sup>2</sup> | | | | |

Statistical Analysis Plan: SAINT

| | T | | 1 | 1 |
|---------------------------------------------------|---|-----|-----|---|
| Troponin T (in ng/mL) <sup>2</sup> | | | | |
| Procalcitonin (in ng/mL) <sup>2</sup> | | | | |
| Sodium (in mEq/L) <sup>2</sup> | | | | |
| Potassium (in mEq/L) <sup>2</sup> | | | | |
| Chlorine (in mEq/L) <sup>2</sup> | | | | |
| Bicarbonate (in mEq/L) <sup>2</sup> | | | | |
| Remaining anion (in mEq/L) <sup>2</sup> | | | | |
| Ferritin (in ng/mL) <sup>2</sup> | | | | |
| CPK (in UI/L) <sup>2</sup> | | | | |
| D-Dimer (in ng/mL) <sup>2</sup> | | | | |
| IL-6 (in pg/mL) <sup>2</sup> | | | | |
| Hemogram | | | | |
| Red blood cells (in 10 <sup>12</sup> /L) | | | | |
| Haemoglobin (in g/dL) | | | | |
| Hto (in %) | | | | |
| VCM (in f/L) | | | | 1 |
| HCM (in pg) | | | | 1 |
| CMHC (in g/dL) | | | | 1 |
| RDW (in %) | | | | 1 |
| Platelets (in 10 <sup>9</sup> /L) | | | | 1 |
| VPM (in f/L) | | | | 1 |
| PWD (in %) | | | | |
| White blood cells (in 10 <sup>9</sup> /L) | | | | |
| Neutrophil (in %) | | | | |
| Neutrophil absolute value (in 10 <sup>9</sup> /L) | | | | 1 |
| Lymphocyte (in %) | | | | |
| Lymphocyte absolute value (in 109/L) | | | | |
| Monocytes (in %) | | | | |
| Monocytes absolute value (in 10 <sup>9</sup> /L) | | | | 1 |
| Eosinophil (in %) | | | | |
| Eosinophil absolute value (in 10 <sup>9</sup> /L) | | | | 1 |
| Basophiles (in %) | | | | 1 |
| Basophiles absolute value (in 10 <sup>9</sup> /L) | | | | 1 |
| Platelet-Lymphocyte index | | | | 1 |
| Neutrophil-Lymphocyte index | | | | 1 |
| Severity predictor?? (N/L*CRP*D-dimer) | | | | |
| 1: n/N (Percentage) | 1 | II. | II. | 1 |

- 1: n/N (Percentage)
- 2: Median (IQR) [n]
- 3: includes General malaise, Myalgia, Appetite, Headache
- 4: ENT: Ear, Nose, Throat (includes anosmia and dysgeusia)
- 5: only women considered in this section


Statistical Analysis Plan: SAINT

Table 3. PCR positivity

| Variable | Study arm | | RR (95% CI) | p-value <sup>2</sup> |
|---|---|---|---|---|
| Variable | Placebo | Ivermectin | KK (33% CI) | p-value |
| Positive PCR at day 7 <sup>1</sup> | | | | |
| Positive PCR culture at day 4 <sup>1</sup> | | | | |
| Positive PCR culture at day 7 <sup>1</sup> | | | | |

<sup>1:</sup> n/N (Column percentage)

RR: risk ratio, CI: confidence interval

Table 4. Seroconversion at day 21

| Variable | Study | All subjects | |
|---|---|---|---|
| Variable | Placebo | Ivermectin | All subjects |
| Seroconversion at day 21 <sup>1</sup> | | | |

<sup>1:</sup> n/N (Column percentage)

Table 5. Seroconversion at day 21 in patients taking ivermectin

| Variable | PCR at day 7 | |
|---------------------------------------|--------------|----------|
| Valiable | Negative | Positive |
| Seroconversion at day 21 <sup>1</sup> | | |

<sup>1:</sup> n/N (Column percentage)

Table 6. AEs description

| Variable | Stud | All subjects | |
|---|---|---|---|
| variable | Placebo | Ivermectin | All subjects |
| Number of AEs observed | | | |
| Number of SAEs observed | | | |
| Drug-related SAEs <sup>2</sup> | | | |
| Observed serious adverse events (per su | | | |
| Number of SAEs during FU <sup>1</sup> | | | |
| Death <sup>2</sup> | | | |
| Body as a whole <sup>2</sup> | | | |
| Gastrointestinal <sup>2</sup> | | | |
| Nervous System/Psychiatric <sup>2</sup> | | | |
| Skin <sup>2</sup> | | | |

<sup>1:</sup> Median (IQR) [n]

<sup>2:</sup> Fisher's exact test

<sup>2:</sup> n/N (Percentage)

Statistical Analysis Plan: SAINT

**Table 7.** Treatment effect on symptom presence

| Variable | OR (95% CI) | p-value <sup>1</sup> |
|-----------|-------------|----------------------|
| Treatment | | |
| Day | | |

<sup>1:</sup> Mixed effect logistic regression model with subject as a random intercept

## 15.2 Listings

**List 1**. Patient baseline information

| Patient | Study arm | Ct | Vital signs | Symptoms | Lab results + immuno |
|---------|------------|-------|-------------|----------|----------------------|
| 1 | Placebo | value | | | |
| 2 | Placebo | | | | |
| 3 | Placebo | | | | |
| 4 | Placebo | | | | |
| 5 | Placebo | | | | |
| 6 | Placebo | | | | |
| 7 | Placebo | | | | |
| 8 | Placebo | | | | |
| 9 | Placebo | | | | |
| 10 | Placebo | | | | |
| 11 | Placebo | | | | |
| 12 | Placebo | | | | |
| 13 | Ivermectin | | | | |
| 14 | Ivermectin | | | | |
| 15 | Ivermectin | | | | |
| 16 | Ivermectin | | | | |
| 17 | Ivermectin | | | | |
| 18 | Ivermectin | | | | |
| 19 | Ivermectin | | | | |
| 20 | Ivermectin | | | | |
| 21 | Ivermectin | | | | |
| 22 | Ivermectin | | | | |
| 23 | Ivermectin | | | | |
| 24 | Ivermectin | | | | |


Statistical Analysis Plan: SAINT

**List 2**. List of all AEs occurred

| Study arm | AE diagnosis | Drug relatedness | Severity | Action taken | Withdrawal due to AE |
|---|---|---|---|---|---|

#### List 3. List of all SAEs occurred

| Study arm | AE diagnosis | Drug relatedness | Severity | Action taken | Withdrawal due to AE |
|---|---|---|---|---|---|

### 15.3 Figures

Figure 1. Viral load evolution during FU (days 1, 4, 7, 14 and 21) by study arm

This figure will contain a boxplot for each day and study arm.

[boxplots]

Figure 2. Viral load change during FU (days 1, 4, 7, 14 and 21) by study arm

A boxplot for each day and study arm.

[boxplots]

Figure 3. Viral load evolution during FU (days 1, 4, 7, 14 and 21) by study participant

Separate line plots that will show each subject's evolution during FU.

[line plots]

Figure 4. Symptom presence during FU (days 1, 4, 7, 14 and 21) by study arm

One diagram for each symptom considered: General (General malaise, Myalgia, Appetite, Headache), ENT (includes anosmia and dysgeusia), Respiratory and Digestive.

[Alluvial diagram]

Statistical Analysis Plan: SAINT

Figure 5. System abnormalities identified during FU (days 1, 4, 7, 14 and 21) by study arm

One diagram for each system considered: General Appearance, Heart, Lungs, Abdomen and Extremities.

[Alluvial diagram]

Figure 6. Time to symptom improvement by study arm

One graph for the composite outcome "any symptom" and one for each symptom considered: General (General malaise, Myalgia, Appetite, Headache), ENT (includes anosmia and dysgeusia), Respiratory and Digestive.

[Kaplan-Meier curve]

Figure 7. Time to severe disease or death by study arm

[Kaplan-Meier curve]
